CLINICAL TRIAL: NCT00600860
Title: A Prospective, Multicentre European Registry for Newly Diagnosed Patients With Myelodysplastic Syndromes (MDS), Including Acute Myeloid Leukaemia With 20-<30 Percent Marrow Blasts (Former RAEB-t), and Chronic Myelomonocytic Leukaemia (CMML)
Brief Title: A Prospective, Multicentre European Registry for Newly Diagnosed Patients With Myelodysplastic Syndromes
Acronym: EUMDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 883
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Myelodysplastic Syndromes (MDS)
Keywords: MDS (all IPSS subtypes); Newly diagnosed
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Bone marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MDS patients: Patients with MDS according to current WHO criteria and International Prognostic Scoring System (IPSS) classification
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — Only registration of clinical practice

SUMMARY:
Study Objectives:

To collect and describe demographics, disease-management, and treatment outcomes of Myelodysplastic Syndromes (MDS) patients who are newly diagnosed and classified according to the World Health Organization (WHO) criteria.

To perform observational studies concerning relevant scientific research questions in MDS using clinical data and biological samples, and to present relevant research outcomes in the fields of diagnosis and prognostication, health related quality of life issues, health economics, and risk stratification for newly developed classes of drugs.

To disseminate results of the studies to all stakeholders involved.

DETAILED DESCRIPTION:
Methodology:

Data on patients with MDS will be collected prospectively at diagnosis and at 6-months intervals after diagnosis. The data will be gathered by seventeen (or more) countries that are represented within the LeukemiaNet MDS Working Party and will be combined in one central European Database. Data analyses will be conducted by the Data Management Centre at the University of York in various sub studies, at specific time points as decided or requested by the steering committee, but at least once a year included in the European Registry and at the end of the follow-up period.

Number of Patients & Centres Over 149 hematology centres in eighteen (or more) different countries (Austria, Croatia, Czech Republic, Denmark, France, Germany, Greece, Israel, Italy, The Netherlands, Romania, Spain, Sweden, Switzerland and United Kingdom) will participate as referral centres in this Registry. The recruitment target is a minimum of 3000 cases lower-risk MDS and 1000 higher-risk cases.

Population:

The study population will consist of newly diagnosed patients with all subtypes of MDS classified according to the WHO criteria, including therapy-related MDS and MDS-F, AML with 20-<30 percent marrow blasts (former RAEB-t), and CMML and other forms of mixed MDS/MPD.

Study Duration:

The enrolment time is scheduled to continue until at least December 2022 but extension of the recruitment period is possible. Patients will be followed until withdrawal (for any reason) or termination of the EUMDS Registry.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria

* Age > 18 years
* Newly diagnosed patient (within 100 days from the date of the diagnostic bone marrow (BM) aspirate)
* MDS classified according to current WHO criteria

  * All sub groups of MDS
  * Therapy-related MDS
  * MDS with Fibrosis (MDS-F)
  * AML with 20-<30 percent marrow blasts (former RAEB-t)
  * CMML and other forms of mixed MDS/MPD
* IPSS and IPSS-R Risk group classification (mandatory)
* Able and willing to provide the written informed consent

Exclusion Criteria:

* Age <18 years
* Patient unwilling or unable to give consent
* AML with ≥30 percent marrow blasts according to WHO
* Patients with inv(16), t(5;17) and t(8;21) are considered AML and therefore not eligible
* Patients with higher risk MDS progressed from a previously diagnosed lower risk MDS that was not registered within 100 days after first diagnosis of (lower risk) MDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinic
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2008-04; Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Demographics | 14.5 years of follow-up (FU)
  The primary objective of this study is collect and describe demographics, clinical and lab manifestations, epidemiological data, genetic characteristics, HRQoL, disease-management, and treatment outcomes of MDS patients who are newly diagnosed and classified according to the WHO-2008 and WHO-2016 criteria

SECONDARY OUTCOMES:
Correlations | 14.5 years of FU
  To investigate the relationship between:
  * Clinical characteristics at inclusion and during follow-up
  * Treatments received, including transfusions, and
  * Responses to treatment
  * Overall survival
  * Disease progression
  * General and disease specific HRQoL, and Karnofsky Performance Status
  * Health Economics
New prognostic scoring systems | 14.5 years of FU
  To derive and validate new prognostic scoring systems
Scientific research in MDS | 14.5 years of FU
  To perform observational studies concerning relevant scientific research questions in MDS using clinical data and biological samples and to present relevant research outcomes in the fields of diagnosis & prognostication, HRQoL issues, health economics, risk stratification for newly developed classes of drugs.

OTHER OUTCOMES:
Dissemination | 14.5 years of FU
  To disseminate the results of the studies to all stakeholders involved

CONTACTS AND LOCATIONS:
Overall Officials: David Bowen, PhD, Study Chair — Leeds General Infirmary; Theo de Witte, Prof Dr, Study Director — Radboud University Medical Center
Locations (18):
- University of Innsbruck Fachartz fur Innere Medizin, Dept of Hematology, Innsbruck, Austria
- Clinical Hospital Merkur, Zagreb, Croatia
- Institute of Haematology and Blood Transfusion U nemocnice, Prague, Czechia
- Aarhus University Hospital, Aarhus, Denmark
- Hopital Avicenne Universite Paris, Dept of Hematology, Paris, France
- Medizinische Klinik und Poliklinik fur Haematologie, Onkologie und Klinische Immunologie, Düsseldorf, Germany
- University of Patras Medical School, Haematology Division, Dept of Internal Medicine, Pátrai, Greece
- Tel-Aviv Sourasky Medical Center, Dept. of Medicine A, Tel Aviv, Israel
- University of Pavia Medical SChool, Dept of Hematology, Pavia, Italy
- Radboud University Nijmegen Medical Centre, dept of Hematology, Nijmegen, Netherlands
- Medical University, Dept of Hematology, Oncology and Internal Medicine, Warsaw, Poland
- Instituto Português de Oncologia de Lisboa,, Lisbon, Portugal
- Fundeni CLinical Institute, Clinic of Hematology, Bucharest, Romania
- Clinical Center of Vojvodina, Novi Sad, Serbia
- Hospital La Fe, Dept of Hematology, Valencia, Spain
- Karolinsky Institute Huddinge University Hospital, Dept of Medicine Division HAematology, Stockholm, Sweden
- Inselspital, Bern, Switzerland
- Leeds General Infirmary Dept of Hematology, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The study results (aggregated data) will be published in an academic journal and presented at scientific meetings. We are working on an update of the website: www.eumds.org. EUMDS related activities and results are also shared via www.mds-europe.eu.

REFERENCES:
- [Derived] Garelius HKG, Bagguley T, Taylor A, Fenaux P, Bowen D, Symeonidis A, Mittelmann M, Stauder R, Cermak J, Sanz G, Langemeijer S, Malcovati L, Germing U, Sanhes L, d'Aveni M, Culligan D, Kotsianidis I, Koinig KA, van Marrewijk C, Crouch S, deWitte T, Smith A, Hellstrom-Lindberg E. Survival and quality of life in patients with lower risk myelodysplastic syndromes exposed to erythropoiesis-stimulating agents: an observational cohort study. Lancet Haematol. 2025 Feb;12(2):e128-e137. doi: 10.1016/S2352-3026(24)00350-8. PMID 39909656
- [Derived] Rombaut D, Sandmann S, Tekath T, Crouch S, de Graaf AO, Smith A, Painter D, Kosmider O, Tobiasson M, Lennartsson A, van der Reijden BA, Park S, D'Aveni M, Slama B, Clappier E, Fenaux P, Ades L, van de Loosdrecht A, Langemeijer S, Symeonidis A, Cermak J, Preudhomme C, Savic A, Germing U, Stauder R, Bowen D, van Marrewijk C, Bernard E, de Witte T, Varghese J, Hellstrom-Lindberg E, Dugas M, Martens J, Malcovati L, Jansen JH, Fontenay M; MDS-RIGHT consortium. Somatic mutations and DNA methylation identify a subgroup of poor prognosis within lower-risk myelodysplastic syndromes. Hemasphere. 2025 Jan 22;9(1):e70073. doi: 10.1002/hem3.70073. eCollection 2025 Jan. PMID 39850648
- [Derived] Stojkov I, Conrads-Frank A, Rochau U, Arvandi M, Koinig KA, Schomaker M, Mittelman M, Fenaux P, Bowen D, Sanz GF, Malcovati L, Langemeijer S, Germing U, Madry K, Guerci-Bresler A, Culligan DJ, Kotsianidis I, Sanhes L, Mills J, Puntscher S, Schmid D, van Marrewijk C, Smith A, Efficace F, de Witte T, Stauder R, Siebert U. Determinants of low health-related quality of life in patients with myelodysplastic syndromes: EUMDS Registry study. Blood Adv. 2023 Jun 27;7(12):2772-2783. doi: 10.1182/bloodadvances.2022008360. PMID 36607832
- [Derived] de Swart L, Crouch S, Hoeks M, Smith A, Langemeijer S, Fenaux P, Symeonidis A, Cermak J, Hellstrom-Lindberg E, Stauder R, Sanz G, Mittelman M, Holm MS, Malcovati L, Madry K, Germing U, Tatic A, Savic A, Almeida AM, Gredelj-Simec N, Guerci-Bresler A, Beyne-Rauzy O, Culligan D, Kotsianidis I, Itzykson R, van Marrewijk C, Blijlevens N, Bowen D, de Witte T; EUMDS Registry Participants. Impact of red blood cell transfusion dose density on progression-free survival in patients with lower-risk myelodysplastic syndromes. Haematologica. 2020 Mar;105(3):632-639. doi: 10.3324/haematol.2018.212217. Epub 2019 Jun 6. PMID 31171638
- [Derived] Itzykson R, Crouch S, Travaglino E, Smith A, Symeonidis A, Hellstrom-Lindberg E, Sanz G, Cermak J, Stauder R, Elena C, Germing U, Mittelman M, Langemeijer S, Madry K, Tatic A, Holm MS, Almeida AM, Savic A, Simec NG, Luno E, Culligan D, Guerci-Bresler A, Malcovati L, van Marrewijk C, Bowen D, de Witte T, Fenaux P; European MDS Registry members. Early platelet count kinetics has prognostic value in lower-risk myelodysplastic syndromes. Blood Adv. 2018 Aug 28;2(16):2079-2089. doi: 10.1182/bloodadvances.2018020495. PMID 30126931
- [Derived] de Swart L, Reiniers C, Bagguley T, van Marrewijk C, Bowen D, Hellstrom-Lindberg E, Tatic A, Symeonidis A, Huls G, Cermak J, van de Loosdrecht AA, Garelius H, Culligan D, Macheta M, Spanoudakis M, Panagiotidis P, Krejci M, Blijlevens N, Langemeijer S, Droste J, Swinkels DW, Smith A, de Witte T; EUMDS Steering Committee. Labile plasma iron levels predict survival in patients with lower-risk myelodysplastic syndromes. Haematologica. 2018 Jan;103(1):69-79. doi: 10.3324/haematol.2017.171884. Epub 2017 Nov 9. PMID 29122992
- [Derived] Garelius HK, Johnston WT, Smith AG, Park S, de Swart L, Fenaux P, Symeonidis A, Sanz G, Cermak J, Stauder R, Malcovati L, Mittelman M, van de Loosdrecht AA, van Marrewijk CJ, Bowen D, Crouch S, de Witte TJ, Hellstrom-Lindberg E. Erythropoiesis-stimulating agents significantly delay the onset of a regular transfusion need in nontransfused patients with lower-risk myelodysplastic syndrome. J Intern Med. 2017 Mar;281(3):284-299. doi: 10.1111/joim.12579. Epub 2016 Dec 7. PMID 27926979
- See also: European MDS Registry — http://www.eumds.org
- See also: European MDS network platform — https://mds-europe.eu/
- See also: Publication (PMID: 28526957): Cytomorphology review of 100 newly diagnosed lower-risk MDS patients in the European LeukemiaNet MDS (EUMDS) registry reveals a high inter-observer concordance — https://link.springer.com/article/10.1007%2Fs00277-017-3009-7
- See also: Publication (PMID: 29122992): Labile plasma iron levels predict survival in patients with lower-risk myelodysplastic syndromes — http://www.haematologica.org/content/103/1/69.long
- See also: Publication (PMID: 29572506): Health-related quality of life in lower-risk MDS patients compared with age- and sex-matched reference populations: a European LeukemiaNet study — https://www.nature.com/articles/s41375-018-0089-x
- See also: Publication (PMID: 31171638): Impact of red blood cell transfusion dose density on progression-free survival in lower-risk myelodysplastic syndromes patients — http://www.haematologica.org/content/early/2019/06/05/haematol.2018.212217.long
- See also: Publication (PMID: 31278207): Impact of treatment with iron chelation therapy in patients with lower-risk myelodysplastic syndromes participating in the European MDS registry — http://www.haematologica.org/content/early/2019/07/05/haematol.2018.212332.long